CLINICAL TRIAL: NCT02291328
Title: A Human Intervention Trial Investigating the Effects of Brassica on Gut Lactobacilli
Brief Title: Effects of Brassica on Human Gut Lactobacilli
Acronym: EBL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: The Danish Council for Strategic Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IFR04/2014
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-05

CONDITIONS: Human Gut Microbiota

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Brassica (Experimental): Participants will be asked to consume 3x 84g portions of frozen broccoli, 3x 84g portions of frozen cauliflower, and 3x 300g portions of frozen broccoli and sweet potato soups a week for a total of 2 weeks.
  Interventions: Other: High Brassica
- Low Brassica (Experimental): Participants will be asked to consume 1x 84g portion of either frozen broccoli or frozen cauliflower in week one, and the remaining 84g portion of Brassica in week two.
  Interventions: Other: Low Brassica

INTERVENTIONS:
Other: High Brassica — Participants consume a minimum of one portion of a Brassica food (84g frozen broccoli, 84g frozen cauliflower, or 300g frozen broccoli and sweet potato soup) each day for 14 consecutive days at their homes.
  Arms: High Brassica
Other: Low Brassica — Participants consume one portion of a Brassica vegetable (84g frozen broccoli, or 84g frozen cauliflower) each week for two weeks at their homes.
  Arms: Low Brassica

SUMMARY:
Brassica vegetables are an important part of the investigators normal diet and are associated with a reduced risk of many chronic diseases. The protective effect may be as a result of the hydrolytic products of compounds contained within these vegetables, called glucosinolates. There is evidence that consumption of Brassica vegetables may cause compositional changes to the investigators gut microbiota. The aim of this study is to see whether a diet rich in Brassica alters the human gut microbiota composition, and specifically whether it causes an increase in the number of the beneficial bacteria known as lactobacilli.

DETAILED DESCRIPTION:
The study is a randomised human dietary intervention two-phase cross-over study and will require the participants to consume both a low and a high Brassica vegetable diet. In this study, male and female participants aged between 18 and 50 years will be recruited until 10 complete the study. For the low Brassica diet test phase, the participants will be provided with one 84g portion of frozen broccoli and one 84g portion of frozen cauliflower, to be consumed across a period of two weeks. The participants will be asked to consume one of these portions of Brassica (either broccoli or cauliflower) in week one, and then consume the remaining portion of Brassica in week two, with a minimum of 5 days between consuming the two portions. When on the high Brassica diet test phase, the participants will be provided with six 84g portions of frozen broccoli, six 84g portions of frozen cauliflower, and six 300g portions of frozen broccoli and sweet potato soups (each with a broccoli content of 84g), to be consumed across a period of two weeks. The participants will be asked to consume three portions of broccoli, three portions of cauliflower, and three portions of the broccoli and sweet potato soups each week for two weeks, consuming a minimum of one portion per day. The Brassica diet test phases will be separated by a washout period, which will be a minimum of 2 weeks.

The participants will be asked to restrict their diet of Brassica vegetables and ITC-containing foods for a period which includes 2 weeks prior to test phases 1 and 2, as well as during the full 2 weeks of each test phase. The participants will be asked to provide faecal samples, urine samples, complete food diaries and stool charts at various stages throughout the intervention. Participants will be asked to complete a food diary, recording the consumption of all fruits and vegetables, for a consecutive seven day period, during each of the two test phases (test phases 1 and 2), and for the entire seven days of the last week of the study when consuming their habitual diet. Participants will also need to be willing to complete stool charts noting the frequency and consistency of their bowel movements.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 50.
* Smokers and non-smokers.
* Those with a body mass index (BMI) between 19.5 and 30 kg/m2.
* Those that live within a 40 mile radius of Norwich.

Exclusion Criteria:

* Women who are or have been pregnant within the last 12 months, or are lactating and/or breast feeding.
* Those currently suffering from, or have ever suffered from, any diagnosed gastrointestinal disease, gastrointestinal disorders including regular diarrhoea and constipation (excluding hiatus hernia unless symptomatic) and/or have undergone gastrointestinal surgery, or the study intervention/procedure is contraindicated.
* Have been diagnosed with any long-term medical condition that may affect the study outcome (e.g. diabetes, haemophilia, cardiovascular disease, glaucoma, anaemia). These will be assessed on an individual basis.
* Those diagnosed with a long-term medical condition requiring medication that may affect the study outcome.
* Those regularly taking self-prescribed over the counter medications for digestive/gastrointestinal conditions.
* Those on long-term antibiotic therapy. Those who have been on a course of antibiotics are able to participate in/continue on the study once 4 weeks has elapsed from the end of the course of antibiotics. This will be assessed on an individual basis.
* Those regularly taking laxatives (once a month or more).
* Those intermittently using pre &/or probiotics unless willing to abstain for 1 month prior to and during study period. (If used regularly (3+ times a week, and for more than one month) and will continue throughout study period then do not exclude).
* Those on a diet programme or those who plan to start a diet programme during the study that may affect the study outcome (e.g. the 5:2 fasting diet) unless willing to abstain for 1 month prior to and during study period. These will be assessed on an individual basis.
* Those taking dietary supplements or herbal remedies (including those derived from Brassica plants) which may affect the study outcome - unless the participant is willing to discontinue taking them for 1 month prior to and during study period. Please note that some supplements may not affect the study and this will be assessed on an individual basis.
* Regular/recent (within 3 months) use of colonic irrigation or other bowel cleansing techniques.
* Recently returned to the United Kingdom (UK) following a period abroad, and who have suffered gastric symptoms during the period abroad or on return to the UK. These will be assessed on an individual basis.
* Parallel participation in another research project which involves dietary intervention and/or sampling of biological fluids/materials. Sampling of certain biological samples, such as saliva, may not affect the study and this will be assessed on an individual basis.
* Those who record blood in their stools or have two or more episodes of type 1, 2, or 7 stools during the study.
* Any person related to or living with any member of the study team.
* Those who are unwilling to provide the contact details of their general practitioners (GPs).
* Those who are unable to provide written informed consent.
* Those who are not suitable to take part in this study because of their eligibility screening results.
* Those who do not have access to a freezer.
* Those who regularly consume more than 15 units of alcohol (women) or 22 units of alcohol (men) a week.
* Those who are allergic to any of the foods/ingredients within the foods supplied.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Lactobacilli in human faecal microbiota | Two weeks
  To investigate whether eating a diet rich in Brassica vegetables for two weeks will cause an increase in human gut lactobacilli, compared to the number of lactobacilli present in the participants' normal gut microbiota.

SECONDARY OUTCOMES:
Human faecal microbial community composition | Two weeks
  To ascertain whether eating a diet rich in Brassica vegetables modulates the gut microbial community as a whole, as compared to the consumption of a low Brassica diet, and the participants' normal gut microbiota.
Human faecal bile acid profile | Two weeks
  To determine whether the consumption of a high and/or low Brassica vegetable diet causes a change in short chain fatty acids and bile acids in the faeces.
Faecal bacterial gene expression | Two weeks
  To determine whether the consumption of a high and/or low Brassica vegetable diet causes a change in bacterial gene expression in the faeces.
Urinary isothiocyanates (ITCs) excretion | Two weeks
  To determine the extent of glucosinolate conversion to ITCs from Brassica vegetables, as measured by ITC excretion in the urine.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Mithen, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Institute of Food Research, Norwich, Norfolk, United Kingdom